CLINICAL TRIAL: NCT07312916
Title: Effect of Hand Massage on Chronic Kidney Disease Associated Pruritus in Patients Receiving Hemodialysis: a Mixed Methods Study
Brief Title: Effect of Hand Massage on Chronic Kidney Disease Associated Pruritus in Patients Receiving Hemodialysis
Acronym: MADRID
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Applied Sciences of Western Switzerland (Other)
Collaborators: Swiss National Science Foundation (Other)
Responsible Party: Principal Investigator, Nancy Helou, Full Professour UAS, University of Applied Sciences of Western Switzerland
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 131465
Record Dates: First submitted 2025-12-17; First posted 2025-12-31 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Chronic Kidney Disease Associated Pruritus

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hand-massage (Experimental): Participants randomized to the intervention group (n=27) will receive hand-massage that consists of 10 min hand-massage, two times/week for the first month, then once/week for the two consecutive months, at any time during the hemodialysis session.
  Interventions: Other: Hand-massage
- Control (No Intervention): Participants assigned to the control group (n=27) will receive uninterrupted attention from the nurse via a conversation without use of physical touch for 10 min, two times /week for the first month, then once/month for the two consecutive months, at any time during the hemodialysis session

INTERVENTIONS:
Other: Hand-massage — Hand-massage involves engagement with the patient using an enveloping contact on the whole hand and the forearm by means of rhythmic and circular movements, followed by an application of a hand cream or essential oil to the patient's forearm, wrist, palm and back of hand, and fingers using the same movements. The massage applies moderate pressure to the forearm, light gestures on the wrist and the back of the hand, and moderate pressure on the palm and fingers. It ends with a gradual slowing of the manipulations
  Arms: Hand-massage

SUMMARY:
Chronic Kidney Disease-Associated Pruritus (CKD-aP) affects about 25% of Swiss hemodialysis patients, most with moderate to severe itching. It negatively impacts sleep, quality of life, and survival. This mixed-methods study will investigate the effect hand massage delivered by nurses on the itch severity, health-related quality of life and sleep compared to usual care in patients on hemodialysis. Fifty-four patients will be randomized to receive either hand massage or verbal attention over three months. Quantitative data (VAS, 5D Itch Scale, SF-12, MOS Sleep Scale-R) will be collected at baseline, one, and three months. Qualitative interviews with 12 participants who received the hand massage intervention, will explore their experiences. The intervention is safe, non-invasive, and may offer valuable insights into CKD-aP management and pathogenesis.

DETAILED DESCRIPTION:
Chronic Kidney Disease Associated Pruritus (CKD-aP) represents a distressing skin itch symptom that affects 20-42% of adults on dialysis. We recently conducted the first CKD-aP prevalence study in Switzerland. Results showed that 25% of individuals on hemodialysis experience CKD-aP with 80% suffering from moderate to severe itching. CKD-aP is associated with sleep disturbances, compromised quality of life, social isolation and increased risk of hospitalization and death. CKD-aP may be related to increased uremic toxins, endogenous opioid or immune system dysregulation, peripheral neuropathy with abnormal cutaneous innervation and nerve conduction. In this context, the effect of non-pharmacological management approaches like hand massage on nerve conduction, autonomic stress responses and skin inflammation deserve more attention. Few studies have evaluated the effect of short-term massage (3-4 weeks) on CKD-aP and showed improvement on outcomes evaluated 48 hours after the intervention. The study will be offered to all eligible CKD-aP patients; however, a balanced sex distribution is unlikely due to the male predominance in this population.

This study does not present any risks related to physical or psychological harm to participants. Participants will benefit from a promising non-invasive complementary therapy. Additionally, this study may contribute to a better understanding of the CKD-aP pathogenesis.

The primary objective of this study is to determine whether hand-massage by nurses has an effect on itch severity, Health Related Quality of Life (HRQoL) and sleep in hemodialysis patients with CKD-aP, at one and three months, as compared to usual care, and to explore the lived experience of patients receiving the hand-massage intervention.

A sequential multicenter Explanatory Mixed Methods design will be used. A randomized controlled trial design with two study arms will be conducted first (phase 1), followed by descriptive qualitative research (phase 2).

Phase 1: A total sample size of 54 participants (intervention group n=27; control group n= 27) will be recruted for the RCT. Phase 2: 12 participants from the intervention group who completed the intervention will be recruited to participate in the individual semi-structured interviews.

Participants randomized to the intervention group (n=27) will receive hand-massage that consists of 10 min hand-massage, three times/week for the first month, then once/week for the two consecutive months.

Participants assigned to the control group will receive uninterrupted attention from the nurse via a conversation without use of physical touch for 10 min, three times /week for the first month, then once/month for the two consecutive months.

Questionnaires will be administered by the research assistant who will be blinded to group allocations. Data will be collected at baseline, at one month and at three months, for all outcomes.

Phase 2: Participants from the intervention group who completed the hand-massage intervention will be recruited by the project manager or the research assistant to participate in individual semi-structured interviews.The interviews will be recorded, transcribed and coded using MaxQDA software, enabling a thematic content analysis.

Statistical analyses will be performed in Stata v16 on an intention-to-treat basis. Descriptive statistics will summarize baseline characteristics; between-group differences will be tested with t-tests Repeated measures ANOVA with one between-groups factor (group assignment) and one within-groups factor (time) will be carried out to assess changes in continuous outcome within-subjects across observations. Sex and gender will be recorded and reported in line with HRA/swiss-ethics guidance; subgroup analyses will be explored where numbers allow, acknowledging that balanced sex distribution is unlikely given the epidemiology of the dialysis population.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥18 years
* on hemodialysis ≥ three months
* able to communicate in French
* diagnosed with CKD-aP based on VAS
* signed informed consent

Exclusion Criteria:

* Participants with cognitive impairment -
* participants who have been prescribed CKD-aP medications after enrollment in study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2025-12-17 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Itch severity | at baseline, 1 month, 3 months
  The VAS will also be used to measure CKD-aP severity. It includes two questions. The first refers to the average itch intensity during the last 24h and the second refers to the WI-NRS and addresses the worst itch intensity experienced during the last 24h. VAS score ranges from 0 (not itchy) to 10 (extremely itchy); severity can be classified into five categories: 1) 0 =no itch, 2) 0.1-2.9 points =mild itch, 3) 3.0-6.9 points =moderate itch, 4) 7.0-8.9 points =severe itch, and 5) 9.0-10.0 points =very severe itch
Itch severity and itch related quality of life | at baseline, 1 month, 3 months
  5D itch scale consists of 5-domains (Disability, Distribution, Duration, Degree, and Direction), 5 point-Likert scale designed to measure itch severity and itch-related QoL with an overall score range from 5 to 25. Lower scores indicate less itch severity and a better QoL.
Health related quality of life (HRQoL) | at baseline, 1 month, 3 months
  The Kidney Disease Quality of Life Short Form (KDQOL-SF)™v1.2 questionnaire, a SF-36 derived short-form will be used to measure HRQoL. It is a self-administered 12-question survey assessing eight domains of physical (limitations in physical activities because of health problems, in social activities because of physical or emotional problems, in usual role activities because of physical health problems, bodily pain), and mental health (psychological distress and well-being, limitations in usual role activities because of emotional problems, vitality, and general health perceptions. Scores range between 0-100 and higher scores indicate better HRQoL.
Sleep quality | at baseline, 1 month, 3 months
  Sleep quality will be assessed using the Kidney Disease Quality of Life Short form (KDQOL-SF)™v1.2 Sleep Subscale, composed of four items evaluating sleep quality, difficulty falling asleep, waking up during the night, and feeling rested upon waking. Scores for each item are transformed to a 0-100 scale, with higher scores indicating better sleep quality.

CONTACTS AND LOCATIONS:
Locations (1):
- Etablissements hospitaliers du Nord Vaudois - Hôoital d'Yverdon-les-Bains eHnv, Yverdon-les-Bains, Canton of Vaud, Switzerland

IPD SHARING:
Plan to Share IPD: No